CLINICAL TRIAL: NCT02379143
Title: A Probe Into Practice of the Short Wave Diathermy (SWD) Application in Private Physiotherapy Clinics: a Survey From Ethical Practice & Safety Perspective.
Brief Title: Practice of the Short Wave Diathermy (SWD) Application
Status: Completed | Type: Observational
Sponsor: TPCT's Terna College of Physiotherapy (Other)
Responsible Party: Principal Investigator, DR. SWATI MESHRAM, ASSO. PROF, TPCT's Terna College of Physiotherapy
Other Study IDs: 1
Record Dates: First submitted 2015-02-19; First posted 2015-03-04 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2015-02

CONDITIONS: Electromagnetic Fields
Keywords: SWD, EPA, SAFE PRACTICE

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: interview method: self report form — the responses about participants perception, behavior pattern and attitude were recorded on the self report form

SUMMARY:
Various national & international bodies like FDA, CSP has laid down the guidelines for the reasonable use of SWD electro therapeutic agent (EPA) ensuring safety & effectiveness.

However, it remains uncertain, whether the practicing physiotherapists are aware of the very existence of this guidelines and implementing them in daily practice. Any lack of knowledge about this background can endanger the patient safety leading to serious health hazards.

In the present survey, 49 physiotherapy practitioners were interviewed with a self-report measure to investigate their knowledge base, mode of application of SWD (6 items) & the awareness about recommended guidelines (5 items) etc.

DETAILED DESCRIPTION:
Study design: cross sectional survey design with the use of a self-report form to record the participant's views was used. Sampling frame consisted of physiotherapists working in private clinics in sub-urban area of Mumbai, Maharashtra, India.

Institutional ethic committee of Terna Physiotherapy College granted permission to conduct this survey. The self-report forms were coded in order to conceal the identity of the therapist.

In this survey 49 physiotherapists were interviewed with a self-report form consisting of total 23 item. In the initial section of this survey form a general information was collected regarding years of experience (1 item), Types of condition treated (1 item), No of patients treated (item 1) Duration of onset (item 1) & the type of modality used (item 1). Specific items interrogating therapist's knowledge about the EMF generating modality were designed to retrieve the information about dosage prescription (7 item), acquaintance with recommended guidelines & indications (item 5), years of experience with that particular modality (item1), Any kind of side effects observed (item 1), any action taken for the same (item 2), referring personnel for recommending this modality (item 1), overall therapist's experience with the effectiveness of this modality (item1).

ELIGIBILITY:
Inclusion Criteria:

* Private physical therapists practitioners

Exclusion Criteria:

* Who were volunteering to participate

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 49 PRACTICING PHYSICAL THERAPIST IN PRIVATE CLINICS
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2013-09; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
SELF REPORT FORM | ONE DAY. 15 MINUTES
  This 23 item form was prepared after the extensive discussion with the panel of experts. In the initial section of this survey form a general information was collected regarding years of experience (1 item), Types of condition treated (1 item), No of patients treated (item 1) Duration of onset (item 1) & the type of modality used (item 1). Specific items interrogating therapist's knowledge about the EMF generating modality were designed to retrieve the information about dosage prescription (7 item), acquaintance with recommended guidelines & indications (item 5), years of experience with that particular modality (item1), Any kind of side effects observed (item 1), any action taken for the same (item 2), referring personnel for recommending this modality (item 1), overall therapist's experience with the effectiveness of this modality (item1).

REFERENCES:
- [Result] Bibliography: 1. William E. Prentice PD P, ATC, Professor. Therapeutic Modalities for Physical Therapists. University of North Carolina Chapel Hill, North Carolina. : McGraw-Hill Medical,medical publishing division; 2001. 576 p. 2. Bioelectronics Corporation.